CLINICAL TRIAL: NCT03998462
Title: Mindfulness Based Stress Reduction for Parkinson's Disease: A Longitudinal Study
Acronym: MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3154-R
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
Keywords: Mindfulness; Parkinson's disease; Intervention; Mindfulness Based Stress Reduction (MBSR); Mood; Cognition; Quality of Life
MeSH Terms: conditions — Parkinson Disease | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Assessor are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Based Stress Reduction (MBSR) (Active Comparator): Individuals with Parkinson's disease were randomly assigned to one of two study arms: MBSR or PSC. The MBSR intervention was based on the standard program developed by Jon Kabat-Zinn (1990). It consisted of weekly 2.5 hours sessions x 8 weeks and one 4-hour retreat during week 7. Due to the COVID-19 pandemic, all MBSR sessions were conducted completely online with randomized groups of 6-9 individuals with PD and were led by a trained instructor who was not involved in the clinical care or assessment of the participants.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Psychoeducational Supportive Care (PSC) (Active Comparator): Individuals with Parkinson's disease were randomly assigned to one of two study arms: MBSR or PSC. PSC is a novel intervention developed by Schiehser and colleagues to serve as a control for MBSR in this trial. PSC was modeled after common support/education groups that provide support and psychoeducation about Parkinson's disease available in the community. PSC consisted of weekly 2.5 hours sessions x 8 weeks and one 4-hour "retreat" during week 7. Due to the COVID-19 pandemic, all sessions were conducted completely online with randomized groups of 6-9 individuals with PD and were led by a trained instructor who was not involved in the clinical care or assessment of the participants.
  Interventions: Behavioral: Psychoeducational Supportive Care

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — MBSR used in this trial was based on the standard program developed by Jon Kabat-Zinn (1990). It consisted of weekly 2.5 hours sessions x 8 weeks and one 4-hour retreat during week 7. Due to the COVID-19 pandemic, the MBSR sessions were conducted completely online with randomized groups of 6-9 individuals with PD and were led by a trained instructor who was not involved in the clinical care or assessment of the participants.
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction (MBSR)
Behavioral: Psychoeducational Supportive Care — PSC is a novel intervention developed by Schiehser and colleagues to provide psychoeducation about Parkinson's disease and supportive group care. PSC consisted of weekly 2.5 hours sessions x 8 weeks and one 4-hour "retreat" during week 7. Due to the COVID-19 pandemic, all sessions were conducted completely online with randomized groups of 6-9 individuals with PD and were led by a trained instructor who was not involved in the clinical care or assessment of the participants.
  Other Names: PSC
  Arms: Psychoeducational Supportive Care (PSC)

SUMMARY:
To investigate the efficacy of Mindfulness-based Stress Reduction (MBSR) to improve quality of life, cognition, and mood, as well as to determine the longevity of the treatment response in individuals with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Eligible study participants with PD were randomly assigned to one of two 9-week remote (online) interventions: 1) Mindfulness Based Stress Reduction (MBSR) or 2) Psychoeducational Supportive Care (PSC). Intervention groups consisted of approximately 6-9 individuals and met weekly for 2.5 hours x 8 weeks and for 4 hours ("retreat") during week 7. All participants were remotely administered a battery of neuropsychological tests to measure quality of life, cognition (e.g., executive function, attention, memory), and mood (i.e., anxiety, depression, and apathy), as well as motor symptoms, disease severity, and mindfulness engagement/practice at pre-intervention (baseline), post-intervention (9 weeks), and at 6- and 12-months (follow-up assessments).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of PD based on UK Brain Bank Criteria
2. 40 years of age or older

Exclusion Criteria:

1. Secondary causes of Parkinsonism (e.g. corticobasal degeneration, progressive supranuclear palsy, drug-induced parkinsonism)
2. Other neurological conditions (e.g. stroke)
3. Clinical diagnosis of dementia based on any previous neuropsychological testing
4. Psychosis, antipsychotic treatment or treatment for substance abuse
5. Uncorrected vision or hearing to adequately participate in the intervention
6. Prior formal training in MBSR or regular current MBSR practice
7. Inability to use a computer or technology for participation
8. Active/current suicidal ideation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M. Schiehser, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Psychoeducational Supportive Care (PSC)
Started | 52 | 51
Completed | 40 | 45
Not Completed | 12 | 6
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Technical Difficulties | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Psychoeducational Supportive Care (PSC) | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (7.44) | 69.8 (8.3) | 68.98 (7.895)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 29 | 31 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Non-Hispanic vs. Hispanic
  Participants
    Ethnicity: Non-Hispanic | 46 | 48 | 94
    Ethnicity: Hispanic | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Parkinson's Disease Questionnaire-39
Description: Parkinson's disease Quality of Life (PDQ-39); Total Score = 0-156; higher score = worse quality of life.
Time Frame: pre- to post-intervention (0 to 9 weeks)
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Psychoeducational Supportive Care (PSC)
Number analyzed (Participants) | 52 | 51
change score | -1.03 (9.71) | -3.04 (7.94)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction (MBSR) vs Psychoeducational Supportive Care (PSC); Test type: Superiority; p = 0.34, Mixed Models Analysis; Mean Difference (Final Values) = 1.85, Standard Error of Mean 1.92

2. Secondary Outcome: Matrix Reasoning Test
Description: Test My Brain (TMB) Matrix Reasoning Test (MRT); Total Score = 0-36; higher score = better performance.
Time Frame: pre- to post-intervention (0 to 9 weeks)
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Psychoeducational Supportive Care (PSC)
Number analyzed (Participants) | 52 | 51
change score | 0.154 (6.54) | 1.04 (5.92)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction (MBSR) vs Psychoeducational Supportive Care (PSC); Test type: Superiority; p = 0.41, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, Standard Error of Mean 1.25

3. Secondary Outcome: State-Trait Anxiety Inventory
Description: State-Trait Anxiety Inventory - Trait Subscale (STAI-Trait); 20-80; higher score = higher levels of anxiety.
Time Frame: pre- to post-intervention (0 to 9 weeks)
Measure: Mean (Standard Deviation); unit: change score
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Psychoeducational Supportive Care (PSC)
Number analyzed (Participants) | 52 | 51
change score | -1.40 (4.51) | -1.84 (5.28)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction (MBSR) vs Psychoeducational Supportive Care (PSC); Test type: Superiority; p = 0.71, Mixed Models Analysis; Mean Difference (Final Values) = 0.398, Standard Error of Mean 1.05

ADVERSE EVENTS:
Time Frame: during intervention (~9 weeks)
Arm/Group | Mindfulness Based Stress Reduction (MBSR) | Psychoeducational Supportive Care (PSC)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/52 | 1/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (MBSR) (N=52) | Psychoeducational Supportive Care (PSC) (N=51)
injury during session while performing unprescribed exercise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant injured ribs while performing unprescribed exercise/advanced movement during intervention session. Was evaluated at urgent care and released. Participant fully recovered and resumed future intervention sessions without incident.

LIMITATIONS AND CAVEATS:
Outcome measures were adjusted and/or modified in order to be administered online due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT03998462/Prot_SAP_000.pdf